CLINICAL TRIAL: NCT05225051
Title: N-homocysteinylated Huntingtin in Huntington's Disease
Brief Title: N- Homocysteinylated Huntingtin in Huntington's Disease
Acronym: HO-HD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENAUD Mathilde, Principal Investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-A00407-34
Record Dates: First submitted 2022-01-11; First posted 2022-02-04 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Huntington Disease
Keywords: homocysteinemia
MeSH Terms: conditions — Huntington Disease; Homocysteinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- presymptomatic HD individuals with UHDRS motor ≤ 5 (Mutated Huntingtin) (Experimental): presymptomatic HD individuals with UHDRS motor ≤ 5 (Mutated Huntingtin)
  Interventions: Other: skin biopsy
- symptomatic HD individuals with motor UHDRS > 5 (Mutated Huntingtin) (Experimental): symptomatic HD individuals with motor UHDRS > 5 (Mutated Huntingtin)
  Interventions: Other: skin biopsy
- human control cell lines, Unmutated Huntingtin (Experimental): human control cell lines, Unmutated Huntingtin
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy — skin biopsy

SUMMARY:
Descriptive analysis of N- homocysteinylated Huntingtin in 3 groups of human fibroblasts:

1. presymptomatic HD individuals with UHDRS motor ≤ 5 (Mutated Huntingtin),
2. symptomatic HD individuals with motor UHDRS > 5 (Mutated Huntingtin)
3. human control cell lines, unmutated Huntingtin

DETAILED DESCRIPTION:
Prospective inclusions of 32 subjects with 24 symptomatic HD patients and 8 presymptomatic HD patients.Rationale: This is a pilot study in humans. Over a period of 2 years, the potential recruitment should make it possible to include 32 patients This number will make it possible to calculate the overall variability of the dosage and to have statistics of position and dispersion in the 2 subgroups identified.

Controls: Eight standardized cell lines from human fibroblasts

ELIGIBILITY:
Inclusion Criteria:

* Patient with the symptomatic or presymptomatic Huntington's disease gene (CAG >= 36)
* Molecularly confirmed Huntington's disease
* Patient 18 years of age and older
* Person affiliated to or benefiting from a social security assurance

Exclusion Criteria:

* Person deprived of liberty by a judicial or administrative decision, persons subject to psychiatric care pursuant to Articles L. 3212-1 and L. 3213-1
* Pregnant woman, parturient or nursing mother
* Women of childbearing potential who do not have effective contraception
* Intellectual deterioration preventing the understanding of research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Huntingtin homocysteinylated level | Through study completion, an average of 2 years
  measures the interaction between Homocysteine and Huntingtin in fibroblasts

SECONDARY OUTCOMES:
Blood levels of B9, B12 | Through study completion, an average of 2 years
  Blood levels of B9, B12
Blood levels of homocysteinemia | Through study completion, an average of 2 years
  Blood levels of homocysteinemia

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Renaud, Principal Investigator — CHRU Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Geoffroy A, Kerek R, Pourie G, Helle D, Gueant JL, Daval JL, Bossenmeyer-Pourie C. Late Maternal Folate Supplementation Rescues from Methyl Donor Deficiency-Associated Brain Defects by Restoring Let-7 and miR-34 Pathways. Mol Neurobiol. 2017 Sep;54(7):5017-5033. doi: 10.1007/s12035-016-0035-8. Epub 2016 Aug 17. PMID 27534418
- [Result] Bossenmeyer-Pourie C, Smith AD, Lehmann S, Deramecourt V, Sablonniere B, Camadro JM, Pourie G, Kerek R, Helle D, Umoret R, Gueant-Rodriguez RM, Rigau V, Gabelle A, Sequeira JM, Quadros EV, Daval JL, Gueant JL. N-homocysteinylation of tau and MAP1 is increased in autopsy specimens of Alzheimer's disease and vascular dementia. J Pathol. 2019 Jul;248(3):291-303. doi: 10.1002/path.5254. Epub 2019 Mar 19. PMID 30734924